CLINICAL TRIAL: NCT05408325
Title: Serum Levels of Intercellular Adhesion Molecule-1 and TNF-α in Patients With COVID-19 and Its Relation to Disease Severity
Brief Title: Intercellular Adhesion Molecule-1 and TNF-α in Patients With COVID-19
Status: Completed | Type: Observational
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, AMIRA HUSSEIN ALLAM, assistant professor of chest diseases and tuberculosis, Benha University
Other Study IDs: TEJB-D-22-00066
Record Dates: First submitted 2022-06-04; First posted 2022-06-07 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; Cytokine Storm
Keywords: Covid19; ICAM; Cytokines; TNF
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- confirmed COVID 19 ptients: All patients confirmed by RT-PCR, as positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) who visited the emergency room and the outpatient clinic in the study period.
- healthy subjects: normal healthy volunteers

SUMMARY:
This study aimed to assess the cytokine profile in COVID 19 patients and its relation with disease progression & severity using COVID reporting and data system (CORADS) score.

DETAILED DESCRIPTION:
Study Participants This was a prospective case control study done from February to December 2021, 50 COVID19 patients and 50 control participants after taking their written consents were recruited from the emergency department and outpatient clinic to the Medical microbiology and immunology department and infection control unit in Benha university hospital, Benha, Egypt.

Blood samples were taken at admission from each patient and repeated during the convalescence period for severe pneumonic cases. Serum C-reaction protein (CRP), D-dimer, lipids and glucose were determined by conventional laboratory methods. Blood samples of the control group were also collected and tested. The obtained blood samples were placed in tubes containing EDTA and blank tubes then immediately centrifuged at 1500g and stored at -80°C.

Enzyme-Linked Immunosorbent Assay Quantitative detection for tumor necrosis factor alfa (TNF-α) & intercellular adhesion molecule1 (ICAM-1) was performed using ELISA kits ( Bio reader by thermo fisher scientific Waltham, MA USA) according to the manufacture instructions.

Statistical analysis Data were analysed using SPSS software, version 25.0 (IBM, Armonk, NY, USA) for Windows. Quantitative data were tested for normality using Kolomograph test assuming normality at P>0.05. they were proved to be non parametric, so they were presented as median and inter-quartile range (IQR), and analyzed by Man Whitney U test and Kruskal Wallis (KW) test for independent groups. P ≤0.05 was considered significant

P value >0.05 insignificant P≤0.05 significant P<0.001 highly significant

ELIGIBILITY:
Inclusion Criteria:All patients confirmed by RT-PCR, as positive for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) who visited the emergency room and the outpatient clinic in the study period. The control group included 50 healthy volunteers.

-

Exclusion Criteria:

-

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mild pneumonia was confirmed by positive (qRT-PCR) tests, with no chest tomography features of viral pneumonia, moderate cases had pneumonia in CT chest while severe pneumonia was diagnosed as pneumonia plus 1 of these criteria: (1) respiratory rate ≥ 30 breath per minute with respiratory distress ;(2) saturation of oxygen ≤ 92 % at rest; (3) index of oxygenation ≤ 300 mmHg; (4) respiratory failure that require ventilation;(5) shock; and(6) admission to the ICU unit for other organ failure. CORAD score was calculated for all cases and was included in the radiology report. The degree of suspicion ranged from very low to very high (CO-RADS categories 1-5), while category 0 reflects negative infection and category 6 establishes RT-PCR-positive SARS-Cov-2 infection at time of examination 13.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-02-12 (Actual)

PRIMARY OUTCOMES:
Measure level of ICAM 1 and TNFα in RT PCR positive COVID 19 patients | 12 month
  Quantitative detection for tumor necrosis factor alfa (TNF-α) & intercellular adhesion molecule1 (ICAM-1) was performed using ELISA kits ( Bio reader by thermo fisher scientific Waltham, MA USA) according to the manufacture instructions.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University hospital, Banhā, Kalyobia, Egypt